CLINICAL TRIAL: NCT03119675
Title: Prospective Evaluation of a Smartphone Application, GoCheckKids™ as a Photo Screening Tool in a Pediatric Population
Brief Title: Evaluation of a Smartphone Application, GoCheckKids™ as a Photo Screening Tool in a Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gobiquity Mobile Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-001
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Amblyopia
Keywords: Myopia; Hyperopia; Anisometropia; Amblyopia Risk Factors; Risk Factors; Smartphone Application (App); Photoscreening; Vision Screening; Mobile Vision Screening
MeSH Terms: conditions — Amblyopia; Myopia; Hyperopia; Anisometropia; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photorefraction of ages 1 to 6 years (Other): Clinical Validation of GoCheck Kids Smartphone App
  Interventions: Device: GoCheck Kids (iOS); Device: GoCheck Kids (Windows)

INTERVENTIONS:
Device: GoCheck Kids (iOS) — Photorefraction method is used to screen amblyopia risk factors.
Device: GoCheck Kids (Windows) — Photorefraction method is used to screen amblyopia risk factors.

SUMMARY:
Objective: Prospective evaluation of GoCheckKids™, a smartphone application ('App') as a photo screening device in a pediatric population to detect amblyopia risk factors (ARFs)

Method: Photorefraction images are captured using up to 4 different devices with GoCheckKids™ App and patients are evaluated with cycloplegic refraction.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months to 6 years inclusive.
* Informed consent given by parent or legal guardian.

Exclusion Criteria:

* History of ocular surgery and any condition that would preclude the ability of the investigator to obtain a reliable image and measurement

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 358 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of amblyopia risk factors detected by photo refraction | 1 Day
  Identification of risk factors as compared to gold standard cycloplegic refraction

SECONDARY OUTCOMES:
Number of patients with gaze error identified by photo screening | 1 day
  Detection of gaze error compared to cover test examination results

CONTACTS AND LOCATIONS:
Overall Officials: Sean Donahue, MD, PhD, Principal Investigator — Vanderbilt University